CLINICAL TRIAL: NCT05971212
Title: Can a Supportive Sleep-Practitioner-led Intervention Lead to Improved Sleep, Wellbeing and Reduced Medication Prescribing for Children With Neurodevelopmental Disorders and Co-occurring Severe Sleep Difficulties?
Brief Title: Sleep Support for Children With Neurodevelopmental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SCH-2530
Record Dates: First submitted 2023-06-06; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Sleep Hygiene; Sleep Wake Disorders
MeSH Terms: conditions — Sleep Hygiene; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to Sleep Clinic immediately
  Interventions: Behavioral: Behavioural sleep clinic access
- Control (Experimental): Access to Sleep Clinic delayed
  Interventions: Behavioral: Behavioural sleep clinic access

INTERVENTIONS:
Behavioral: Behavioural sleep clinic access — Access to behavioural Sleep Clinic

SUMMARY:
Around 80% of children with neurodevelopmental disorders such as Attention Deficit Hyperactivity Disorder (ADHD) and autism are reported to have significant difficulties with sleep. This may be a problem with settling off to sleep, waking repeatedly in the night, or both.

Often these children will be prescribed a medication called melatonin to help them sleep, but there is no strong evidence of its effectiveness in children, the long-term side effects are not known and prescriptions for this drug cost millions of pounds a year for the NHS. Many children continue to have persistent sleep problems despite taking melatonin. Sleep support programmes delivered by nurses and sleep practitioners are known to be effective and to give parents and young people long-term strategies for promoting sleep without the use of medication. However, sleep support services are not universally funded.

In this feasibility study 76 children with ADHD, autism or other neurodevelopmental disorder who have been prescribed and have been regularly taking melatonin for at least a year but still have severe sleep difficulties will be recruited. The investigators will help to improve the child's sleep with a sleep practitioner support programme and, if possible, reduce the dose of melatonin or stop it completely if it is no longer needed. Using this design, it will be possible to test whether a programme delivered by sleep practitioners will significantly improve sleep for children using a non-medical approach and in turn improve the health and well-being of the child and family and reduce melatonin prescribing, thereby saving NHS resources and the potential for long-term side effects. The study design will be delivered by Sheffield Children's Hospital and supported by parent users, the Sleep Charity and Sheffield CCG. The results will be disseminated widely to local, regional and national groups as well as via social media.

DETAILED DESCRIPTION:
Sleep is a restorative process, fundamental to physical and psychological health. Sleep disturbances including bedtime resistance and night-time awakening occur in 80% children with neurodisability, the most common associations being with Attention Deficit Hyperactivity Disorder (ADHD), Autism, cerebral palsy and syndromes such as Down, Prader-Willi and Angelman syndromes. In a meta-analysis of subjective and objective studies found that ADHD is associated with higher bedtime resistance, sleep-onset difficulty and longer latency, night awakenings, trouble waking up in the morning, sleep-disordered breathing, daytime sleepiness, more shifts between sleep stages, lower sleep efficiency and less sleep time. Anxiety and depression symptoms may have a significant role in the prevalence of sleep difficulties which would be clearly observed in bedtime resistance, sleep anxiety, night time awakenings and sleep onset delay. Thus, teaching children how to develop sleep hygiene and the use of behavioural modification to manage their fears would help children to fall asleep easily and reduce bedtime resistance which therefore would improve sleep quantity and quality.

The impact of sleep disturbance on children's health is wide-ranging with sleep deprivation leading to difficulties with mood, psychosocial problems and a detrimental impact on the child's cognitive ability and learning. Parents of children with sleep difficulties can suffer high levels of stress and anxiety, decreased ability to work or to drive safely, relationship and financial problems. These stresses lead to an increased demand on NHS primary care services and to prescriptions of drugs such as antidepressants. Children with significant sleep difficulties in the UK are often treated with melatonin, a hormone playing a key role in the timing of sleep-wake cycle, despite the findings of a recent systematic review that suggest that evidence does not strongly support its use. The drug is costly to the health service, with individual Clinical Commissioning Groups (CCGs) spending up to £500k per year on prescription charges for this drug alone.

Evidence from sleep clinics delivered in the local authority, NHS and voluntary sectors has shown that an intensive sleep support intervention can be highly effective. A recent retrospective evaluation of a nurse-led sleep support service successfully discharged 63% children without melatonin prescriptions after a median of two face-to face visits and three telephone calls. The proposed study will aim to support children with neurodevelopmental problems taking melatonin for sleep difficulties to develop long-term strategies for promoting sleep and to reduce drug prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Children to be included will fulfil all of the inclusion criteria.

  * Formal diagnosis of ADHD, autism or another neurodevelopmental condition,
  * Age 4-11 years,
  * Severe sleep disturbance (defined as Score of 3 or more on Composite Sleep Disturbance Index),
  * Been taking melatonin to aid sleep onset for more than 12 months

Exclusion Criteria:

* Exclusion Criteria

  * Already accessed a sleep clinic at Sheffield Children's Hospital or The Sleep Charity.
  * English not first language

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Diary | 20 weeks
  7 day sleep diary (parent report)
Actiwatch data | 20 weeks
  Actiwatch worn for a 7 day period
Child Sleep Habits Questionnaire (CSHQ) | 20 weeks
  Child Sleep Habits Questionnaire (CSHQ)
Melatonin Prescription Status | 20 weeks
  Questionnaire (designed by researchers) asking about patient dosage and type of melatonin taken

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | 20 weeks
  Strengths and Difficulties Questionnaire (SDQ)
CHU-9D Quality of Life questionnaire | 20 weeks
  CHU-9D Quality of Life questionnaire
Healthcare Utilisation | 20 weeks
  Questionnaire (designed by researchers) recording how many times patient has accessed healthcare settings/professionals in last year
Parent Wellbeing | 20 weeks
  Warwick- Edinburgh Mental Wellbeing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Heather Elphick, Study Director — Sheffield Children's NHS Trust
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No